CLINICAL TRIAL: NCT02502513
Title: Can Playing Tetris Prevent the Development of Traumatic Intrusions in Mothers Following an Emergency Cesarean Section? A Pilot Study
Brief Title: Prevention of Intrusive Memories and Posttraumatic Stress Symptoms After Emergency Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Lausanne Hospitals (Other); Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Principal Investigator, Antje Horsch, Research psychologist, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 480/2012
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Posttraumatic Stress Disorder; Acute Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Brief computerized intervention (computer game "Tetris") plus usual care in the maternity department and completion of intrusive memory diary
  Interventions: Behavioral: Brief computerized intervention
- Control (No Intervention): Usual care in the maternity department plus completion of intrusive memory diary

INTERVENTIONS:
Behavioral: Brief computerized intervention — Computer game "Tetris"
  Arms: Intervention

SUMMARY:
This pilot study aims to investigate the effects of a brief computerized intervention (the computer game "Tetris") on intrusive memories and other posttraumatic stress symptoms following an emergency cesarean section. Patients who have undergone an emergency cesarian section will be randomly allocated to either the brief computerized intervention or usual care within the first 6 hours following the operation. Participants will be followed up at one week and one month. It is predicted that participants given the brief computerized intervention will develop fewer intrusive memories and less severe clinical symptoms than those who are not. This will inform the potential future development of a simple computerized intervention to prevent distressing psychological symptoms after a traumatic event such as an emergency cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18+ years
* Had emergency caesarean section within the past 6 hours
* Have given birth to a live baby at ≥ 37 weeks gestation

Exclusion Criteria:

* Do not speak French sufficiently well to participate in assessments
* Have established intellectual disability or psychotic illness
* Baby was transferred to intensive care unit after the birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories recorded by participants in an intrusive memory diary in the week after the emergency cesarean section | 1 week following the emergency cesarean section

SECONDARY OUTCOMES:
Posttraumatic Stress Diagnostic Scale (PDS) | 1 month following the emergency cesarean section
Acute Stress Disorder Scale (ASDS) | 1 week following the emergency cesarean section
Hospital Anxiety and Depression Scale (HADS) | 1 week and 1 month following the emergency cesarean section

OTHER OUTCOMES:
Acceptability of Intervention (rating scale) | 1 month following the emergency cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, DClinPsych, Principal Investigator — CHUV
Locations (1):
- Centre Hôpital Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Horsch A, Vial Y, Favrod C, Harari MM, Blackwell SE, Watson P, Iyadurai L, Bonsall MB, Holmes EA. Reducing intrusive traumatic memories after emergency caesarean section: A proof-of-principle randomized controlled study. Behav Res Ther. 2017 Jul;94:36-47. doi: 10.1016/j.brat.2017.03.018. Epub 2017 Apr 6. PMID 28453969
- See also: Study investigating a related computerized intervention after a road traffic accident in a hospital Emergency Department — https://clinicaltrials.gov/ct2/show/NCT02080351